CLINICAL TRIAL: NCT04853966
Title: The Effects of Physical Activity Tele-Counseling Intervention on Physical Activity, Functional Performance, and Quality of Life in Post-COVID-19 Conditions: A Randomized Controlled Trial
Brief Title: The Effects of Physical Activity Tele-Counseling Intervention in Post-COVID-19 Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Zeliha ÇELİK, Principal Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 219
Record Dates: First submitted 2021-04-18; First posted 2021-04-22 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2021-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Counseling group (Experimental)
  Interventions: Behavioral: Physical activity counseling
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Physical activity counseling — Physical activity counseling will be performed using physical activity behavior steps of the transtheoretical model.
  Arms: Counseling group

SUMMARY:
It has been found that physical activity recommendations with telerehabilitation in different disease groups improve the functional capacity, physical activities and mental health of the patients as much as the supervised exercise programs. However, there are no studies in the literature that provide online physical activity counseling in COVID-19 patients, and evaluate the effect of physical activity counseling on physical activity level, quality of life, physical performance, fatigue, kinesophobia, pain, dyspnea, mental health and behavior change levels. For this reason, this study aimed to evaluate the effect of online physical activity counseling on physical activity level, quality of life, physical performance, fatigue, kinesophobia, pain, dyspnea, mental health and behavior change level in COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have suffered COVID-19 and have passed at 3 months after the Polymerase Chain Reaction (PCR) test turned negative
* Volunteering to participate in the research

Exclusion Criteria:

* Having another diagnosed respiratory or cardiac problem
* Having infections during the evaluation
* Having a skeletal-muscular disease that may affect the evaluation results
* Having neurological and psychiatric problems
* Individuals with restrictions that prevent being physically active during the evaluation and counseling program.
* Pregnant individuals

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-04-17 (Actual); Primary Completion 2022-12-17 (Actual); Study Completion 2023-06-08 (Actual)

PRIMARY OUTCOMES:
Physical activity level | seven days
  Physical activity level will be evaluated multi sensor activity monitor for 7 consecutive days.
General Quality of Life | five minutes
  Quality of Life will be evaluated using Short Form-36 (SF-36) Health Survey Questionnaire

SECONDARY OUTCOMES:
Physical performance | ten minutes
  Physical performance will be evaluated using Short Physical Performance Battery
Dyspnea during daily living activities | two minutes
  Dyspnea using Modified Medical Research Council (MMRC) dyspnea scale will be evaluated. Modified Medical Research Council Dyspnea Scale, levels are graded as 0-4, higher scores imply higher dyspnea.
Behaviour change level | five minutes
  Behaviour change level will be evaluated using Exercise Behaviour Change Scale.
General Pain | one minute
  Pain will be evaluated using Visual Analog Scale
Fear of movement | three minutes
  Fear of movement will be evaluated using Tampa Scale of Kinesiophobia
Fatigue | Two minutes
  Fatigue will be evaluated using Fatigue Severity Scale
Mental Health | three minutes
  Mental Health will be evaluated using Mental Health Continuum Short Form

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Emek, Turkey (Türkiye)

REFERENCES:
- [Derived] Celik Z, Kafa N, Guzel NA, Kokturk N. The effects of physical activity tele-counseling intervention on physical activity, functional performance, and quality of life in post-COVID-19 conditions: a randomized controlled trial. Expert Rev Respir Med. 2024 May;18(5):321-331. doi: 10.1080/17476348.2024.2363862. Epub 2024 Jun 11. PMID 38829396